CLINICAL TRIAL: NCT01776775
Title: The Effect of Postoperative Abdominal Binder to Reduce Seroma Formation and Improve Early Clinical Outcome After Incisional Hernia Repair.
Brief Title: The Effect of Postoperative Abdominal Binder to Improve Outcomes After Incisional Hernia Repair
Acronym: INSAB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to lack of finace
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume Christoffersen, M.D, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INSAB
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia | interventions — Trusses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- abdominal binder (Active Comparator): use of postoperative abdominal binder 30 days after the hernia repair
  Interventions: Device: Abdominal binder
- No abdominal binder (No Intervention): No intervention

INTERVENTIONS:
Device: Abdominal binder — The abdominal binder is worn from immediately after the operation and continuously for 7 days and nights. The belts are standard abdominal binders (ostomy belts) from "ETO garments©" with standard height of 22 cm. and five different sizes in width (S, M, L, XL, XXL- depending on waist measure). A fitting will be done for all included patients before the operation by waist measurement according to the recommendation from the company (see below). When applied, the patients are advised to apply the belt in a lying position.
  Other Names: ETO garments©; ostomy belt; trusses; girdle; longuette; abdominal belt
  Arms: abdominal binder

SUMMARY:
Postoperative seroma formation is one of the most common complications after ventral hernia repair with mesh. Although some seromas may not have clinical impact postoperative seroma formation often causes pain and discomfort and may even compromise wound healing. Abdominal binders (also called trusses, girdle, ostomy belt, longuette or abdominal belt) (AB) are commonly used in abdominal and plastic surgery to prevent seroma formation and diminish pain and discomfort after operation. The primary aim of the present study is to investigate the effect of postoperative abdominal binders after laparoscopic incisional hernia repair on postoperative pain, discomfort and quality of life. Secondary, we register seroma formation. A randomized, controlled, investigator-blinded study supplemented with blinded statistical analysis. We include 60 (2x30) incisional hernia repairs. Patients are randomized either to abdominal binder or no abdominal binder (controls). The abdominal binder is worn from immediately after the operation and continuously for 7 days and nights. All patients have a standardized operation with standardized intra- and postoperative medication regimen. Endpoints measurements are clinically detectable seroma formation scored with seroma classification system buý S. Morales-Conde, pain scored with self-registrations with VAS, and quality of life scored with EQ-5D, recurrence and other complications are also registered. Patients are followed until 90 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

* elective, primary and recurrent laparoscopic and open incisional hernia repair hernia with mesh reinforcement
* fascia defects 6-20 cm measured preoperatively by the surgeon at the out-patient clinic
* patients between 18-80 years

Exclusion Criteria:

* expected low compliance (language problems, dementia and abuse etc.)
* fascia defects >20 cm measured at the preoperative clinical examination.
* acute operation
* decompensated liver cirrhosis (Child-Pugh 3-4)
* patients with a stoma
* if a secondary operation is performed during the hernia repair procedure.
* if a patient withdraws his inclusion consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
seroma formation | 30 days postoperatively
  clinically detectable seroma formation

SECONDARY OUTCOMES:
postoperative pain | pain during the postoperative days 1-3, 7, and 30.
  Measured with self-registration VAS scales

OTHER OUTCOMES:
Quality of life | on day 30 and 90 postoperatively
  measured with EQ-5D
postoperative complications, readmittance, and need for general practitioner visits | 30 days postoperatively
  30-day complications will be registered by patient interview and by cross-checking patient files and the Danish national patient registry
Cosmetic result | 3 months postoperatively
  measured with verbal rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bisgaard, DMSc, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark